CLINICAL TRIAL: NCT04234412
Title: Treatment of Osteoarthritic Knee With High Tibial Osteotomy and Implantation of Allogenic Human Umbilical Cord Blood-derived Stem Cells.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uijeongbu St. Mary Hospital (Other)
Responsible Party: Principal Investigator, Seckjung Kim, Professor, Uijeongbu St. Mary Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC19OISI0134
Record Dates: First submitted 2020-01-05; First posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; knee; high tibial osteotomy; umbilical cord blood stem cell; cartilage regeneration
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Masking Description: only case series of the treated patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osteoarthritic knee patients (Experimental): Osteoarthritic Knee of the patients who will be treated wth high tibial osteotomy and implantation of allogenic human umbilical cord blood-derived stem cells.
  Interventions: Procedure: umbilical cord blood stem cell implantation for osteoarthritis treatment

INTERVENTIONS:
Procedure: umbilical cord blood stem cell implantation for osteoarthritis treatment — The arthroscopic procedure is performed in the supine position after spinal anesthesia. Once the chondral lesion is identified through a standard anteromedial and lateral portal, meniscectomy, meniscal repair, and lateral retinacular release are performed if necessary. microfracture is performed using a microfracture awl.
  Once both the unstable cartilage and subchondral bone are removed in the lesion area and the sclerotic bone is peeled slightly by using a burr, hole(s) are created for implantation by using a drill bit(diameter 4; depth: 4mm). After implantation is performed in the hole by injecting the mixture of sodium hyaluronate and hUCB-MSCs, it is trimmed to the height of the surrounding articular surface.

SUMMARY:
The purpose of this study is to evaluate the clinical results after implantation of human umbilical cord blood-derived mesenchymal stem cells(hUCB-MSCs) and High tibia osteotomy in patients with medial compartment osteoarthritis(MCOA) as well as varus deformity of the knee joint.

This study will prospectively evaluate 10 knees after hUCB-MSCs implantation and High Tibial Osteotomy(HTO) in the medial compartment osteoarthritis and varus deformity of the knee joint.

Clinical outcomes will be evaluated using the International Knee Documentation committee(IKDC), Visual analogue scale(VAS), Western Ontario and McMaster Universities Arthritis Index(WOMAC), and patients satisfaction with the surgery.

ELIGIBILITY:
Inclusion Criteria:

* age older than 30 years,
* full-thickness cartilage lesion measuring at least 2 cm2,
* femoro-tibial angle (varus or valgus) 5°< in the mechanical axis

Exclusion Criteria:

* ligament injuries (such as injuries of the anterior cruciate ligament and posterior cruciate ligament),
* metabolic arthritis
* infectious condition
* psychosis
* serious medical illness
* pregnancy

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
International Cartilage Repair Society (ICRS) grade improvement | at 24, 48, 96 weeks after surgery, score changes will be observed.
  over grade 1 should be improved

SECONDARY OUTCOMES:
Visual analogue scale (VAS) | at 24, 48, 96 weeks after surgery, score changes will be observed.
  0-10 score range, lower the better
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | at 24, 48, 96 weeks after surgery, score changes will be observed.
  0-100 score range, lower the better
International Knee Documentation Committee (IKDC score) | at 24, 48, 96 weeks after surgery, score changes will be observed.
  0-100 % range, lower the better

IPD SHARING:
Plan to Share IPD: Undecided
according to patient agreement, this is flexible.

REFERENCES:
- [Derived] Bae BS, Jung JW, Jo GO, Kim SA, Go EJ, Cho ML, Shetty AA, Kim SJ. Treatment of osteoarthritic knee with high tibial osteotomy and allogeneic human umbilical cord blood-derived mesenchymal stem cells combined with hyaluronate hydrogel composite. Stem Cell Res Ther. 2025 Apr 28;16(1):211. doi: 10.1186/s13287-025-04356-9. PMID 40296133